CLINICAL TRIAL: NCT06700447
Title: Protecting Against HIV Vaccine Misinformation With Adolescent Girls and Young Women in South Africa
Acronym: PROTECT
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: University of Cape Town (Other); Boston University (Other); National Institute of Mental Health (NIMH) (NIH); Health Economics and Epidemiology Research Office, University of the Witwatersrand (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 1R01MH132401 (NIH); 1R01MH132401 (NIH)
Record Dates: First submitted 2024-11-07; First posted 2024-11-22 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Misinformation; HIV Vaccine
Keywords: Prevention: Vaccines; Adolescent Girls and Young Women; South Africa; HIV
MeSH Terms: conditions — Communication

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Active Comparator): Participants enrolled in the control group will receive unrelated information on diabetes and nutrition topics of the same length as the inoculation messages. Please see Appendix 6 for an example of how this message will be structured. This will make the control group an attention control group and ensure that findings are not confounded by the intervention group spending more time and attentional resources on participation in the study.
  Interventions: Behavioral: Nutrition information
- Enhanced inoculation message (Other): Participants enrolled in the enhanced inoculation message arm will receive messages that warn them about impending HIV vaccine misinformation and explains why those claims are false or misleading, the messages will be enhanced with insights from behavioural economics see Appendix 5: "Inoculation message with a BE boost" for an example of the inoculation message. As part of the behavioural economics boost, participants may choose to receive a small token (e.g., sticker, badge, bracelet) with a message promoting vaccination as a consistency and commitment prime.
  Interventions: Behavioral: Enhanced inoculation message

INTERVENTIONS:
Behavioral: Enhanced inoculation message — Participants enrolled in the enhanced inoculation message arm will receive messages that warn them about impending HIV vaccine misinformation and explains why those claims are false or misleading, the messages will be enhanced with insights from behavioural economics see Appendix 5: "Inoculation message with a BE boost" for an example of the inoculation message. As part of the behavioural economics boost, participants may choose to receive a small token (e.g., sticker, badge, bracelet) with a message promoting vaccination as a consistency and commitment prime.
  Arms: Enhanced inoculation message
Behavioral: Nutrition information — Participants enrolled in the control group will receive unrelated information on diabetes and nutrition topics of the same length as the inoculation messages. Please see Appendix 6 for an example of how this message will be structured. This will make the control group an attention control group and ensure that findings are not confounded by the intervention group spending more time and attentional resources on participation in the study.
  Arms: Control

SUMMARY:
Adolescent girls and young women (AGYW) between the ages of 15-29 years continue to bear the brunt of Human Immunodeficiency Virus (HIV) infections in South Africa despite progress recorded in prevention and treatment programmes. The ongoing susceptibility of young women to HIV infection and the sub-optimal uptake of prevention options such as Pre-Exposure Prophylaxis (PrEP) that are highly effective creates a need for an HIV vaccine to benefit populations at substantial risk of HIV infection. However, lessons from previous vaccine studies and the recent COVID-19 vaccine have highlighted significant barriers to vaccine uptake, such as widespread misinformation and vaccine hesitancy. These challenges threaten the successful implementation of a future HIV vaccine. Building on these insights, this study will utilise psychological inoculation theory to develop and evaluate HIV vaccine messages among adolescent girls and young women. Primary objective: To compare changes in intentions to receive HIV vaccine following misinformation exposure in groups with and without psychological inoculation and behavioural economics boost.

Secondary objectives: (1) To compare believability and persuasiveness of misinformation claims and motivational threat associated with misinformation in groups with and without psychological inoculation and behavioural economics boost. (2) To explore subgroup effects by relevant sociodemographic and behavioural factors including HIV risk, PrEP history, COVID-19 vaccine history, general vaccine hesitancy, and information avoidance. The investigators will conduct a two-arm randomized controlled trial of 2-3 inoculation messages that address emerging myths and misinformation about the HIV vaccine in South Africa. Participants will be randomly assigned to a control group or an intervention arm: enhanced inoculation message with insights from behavioural economics.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Age 18-29 years
* Self-reported history of sexual activity in the past 12 months
* Self-reported HIV-negative status or unknown HIV status at enrolment
* Willing and able to provide written informed consent
* Able to read and understand English

Exclusion Criteria:

* Unwilling or unable to provide consent for study participation.

Ages: 18 Years to 29 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Female
Enrollment: 2163 (Actual)
Dates: Start 2025-07-24 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
HIV vaccine intention, at the end of the baseline assessment | At the end of the baseline assessment
  Intention to get the HIV vaccine, measured after inoculation intervention and misinformation exposure The intention to get the vaccine will be measured on a 0-10 scale.

SECONDARY OUTCOMES:
HIV vaccine intention, follow-up | 2-4 weeks
  Intention to get the HIV vaccine, measured at follow-up survey following misinformation exposure and intervention. Measured on a 0-10 scale.
Recommend to friends, at the end of the baseline assessment | At the end of the baseline assessment
  Intention to recommend the HIV vaccine to friends, measured at survey baseline following misinformation exposure and intervention. Measured on a 0-10 scale.
Recommend to friends, follow-up | 2-4 weeks
  Intention to recommend the HIV vaccine to friends, measured at follow-up survey following misinformation exposure and intervention, controlling for baseline pre-intervention/exposure intention. Measured on a 0-10 scale.
Credibility of inoculated exposure #1 | At the end of the baseline assessment
  Extent to which the claim is credible, extent to which the claim makes you anxious or nervous about the HIV vaccine, likelihood of your sharing the claim, for both HIV vaccine claims specifically inoculated against and four new claims. All measured on a 1-7 scale
Credibility of inoculated exposure #2 | At the end of the baseline assessment
  Extent to which the claim is credible, extent to which the claim makes you anxious or nervous about the HIV vaccine, likelihood of your sharing the claim, for both HIV vaccine claims specifically inoculated against and four new claims. All measured on a 1-7 scale
Credibility of inoculated exposure #3 | At the end of the baseline assessment
  Extent to which the claim is credible, extent to which the claim makes you anxious or nervous about the HIV vaccine, likelihood of your sharing the claim, for both HIV vaccine claims specifically inoculated against and four new claims. All measured on a 1-7 scale
Credibility of inoculated exposure #4 | At the end of the baseline assessment
  Extent to which the claim is credible, extent to which the claim makes you anxious or nervous about the HIV vaccine, likelihood of your sharing the claim, for both HIV vaccine claims specifically inoculated against and four new claims. All measured on a 1-7 scale
Credibility of inoculated exposure #5 | At the end of the baseline assessment
  Extent to which the claim is credible, extent to which the claim makes you anxious or nervous about the HIV vaccine, likelihood of your sharing the claim, for both HIV vaccine claims specifically inoculated against and four new claims. All measured on a 1-7 scale
Credibility of inoculated exposure #6 | At the end of the baseline assessment
  Extent to which the claim is credible, extent to which the claim makes you anxious or nervous about the HIV vaccine, likelihood of your sharing the claim, for both HIV vaccine claims specifically inoculated against and four new claims. All measured on a 1-7 scale
Anxiousness of inoculated exposure #1 | At the end of the baseline assessment
  Extent to which the claim makes you anxious or nervous about the HIV vaccine for both HIV vaccine claims specifically inoculated against and four new claims. All measured on a 1-7 scale
Anxiousness of inoculated exposure #2 | At the end of the baseline assessment
  Extent to which the claim makes you anxious or nervous about the HIV vaccine for both HIV vaccine claims specifically inoculated against and four new claims. All measured on a 1-7 scale
Anxiousness of inoculated exposure #3 | At the end of the baseline assessment
  Extent to which the claim makes you anxious or nervous about the HIV vaccine for both HIV vaccine claims specifically inoculated against and four new claims. All measured on a 1-7 scale
Anxiousness of inoculated exposure #4 | At the end of the baseline assessment
  Extent to which the claim makes you anxious or nervous about the HIV vaccine for both HIV vaccine claims specifically inoculated against and four new claims. All measured on a 1-7 scale
Anxiousness of inoculated exposure #5 | At the end of the baseline assessment
  Extent to which the claim makes you anxious or nervous about the HIV vaccine for both HIV vaccine claims specifically inoculated against and four new claims. All measured on a 1-7 scale
Anxiousness of inoculated exposure #6 | At the end of the baseline assessment
  Extent to which the claim makes you anxious or nervous about the HIV vaccine for both HIV vaccine claims specifically inoculated against and four new claims. All measured on a 1-7 scale
Shareability of inoculated exposure #1 | At the end of the baseline assessment
  Likelihood of your sharing the claim for both HIV vaccine claims specifically inoculated against and four new claims. All measured on a 1-7 scale
Shareability of inoculated exposure #2 | At the end of the baseline assessment
  Likelihood of your sharing the claim for both HIV vaccine claims specifically inoculated against and four new claims. All measured on a 1-7 scale
Shareability of inoculated exposure #3 | At the end of the baseline assessment
  Likelihood of your sharing the claim for both HIV vaccine claims specifically inoculated against and four new claims. All measured on a 1-7 scale
Shareability of inoculated exposure #4 | At the end of the baseline assessment
  Likelihood of your sharing the claim for both HIV vaccine claims specifically inoculated against and four new claims. All measured on a 1-7 scale
Shareability of inoculated exposure #5 | At the end of the baseline assessment
  Likelihood of your sharing the claim for both HIV vaccine claims specifically inoculated against and four new claims. All measured on a 1-7 scale
Shareability of inoculated exposure #6 | At the end of the baseline assessment
  Likelihood of your sharing the claim for both HIV vaccine claims specifically inoculated against and four new claims. All measured on a 1-7 scale
Credibility of inoculated exposure #1, follow-up | 2-4 weeks
  Extent to which the claim is credible, extent to which the claim makes you anxious or nervous about the HIV vaccine, likelihood of your sharing the claim, for both HIV vaccine claims specifically inoculated against at baseline. Measured at follow-up on a 1-7 scale
Credibility of inoculated exposure #2, follow-up | 2-4 weeks
  Extent to which the claim is credible, extent to which the claim makes you anxious or nervous about the HIV vaccine, likelihood of your sharing the claim, for both HIV vaccine claims specifically inoculated against at baseline. Measured at follow-up on a 1-7 scale
Shareability of inoculated exposure #1, follow-up | 2-4 weeks
  Extent to which the claim is credible, extent to which the claim makes you anxious or nervous about the HIV vaccine, likelihood of your sharing the claim, for both HIV vaccine claims specifically inoculated against at baseline. Measured at follow-up on a 1-7 scale
Shareability of inoculated exposure #2, follow-up | 2-4 weeks
  Extent to which the claim is credible, extent to which the claim makes you anxious or nervous about the HIV vaccine, likelihood of your sharing the claim, for both HIV vaccine claims specifically inoculated against at baseline. Measured at follow-up on a 1-7 scale
Anxiousness of inoculatedexposure #1, follow-up | 2-4 weeks
  Extent to which the claim is credible, extent to which the claim makes you anxious or nervous about the HIV vaccine, likelihood of your sharing the claim, for both HIV vaccine claims specifically inoculated against at baseline. Measured at follow-up on a 1-7 scale
Anxiousness of inoculated exposure #2, follow-up | 2-4 weeks
  Extent to which the claim is credible, extent to which the claim makes you anxious or nervous about the HIV vaccine, likelihood of your sharing the claim, for both HIV vaccine claims specifically inoculated against at baseline. Measured at follow-up on a 1-7 scale
Credibility of new claims, exposure #7, follow-up | 2-4 weeks
  Extent to which the claim is credible, extent to which the claim makes you anxious or nervous about the HIV vaccine, likelihood of your sharing the claim, for both HIV vaccine claims specifically inoculated against at baseline. Each measured at follow-up on a 1-7 scale for each of 5 claims, and then summed for a global index (range: 5-35).
Credibility of new claims, exposure #8, follow-up | 2-4 weeks
  Extent to which the claim is credible, extent to which the claim makes you anxious or nervous about the HIV vaccine, likelihood of your sharing the claim, for both HIV vaccine claims specifically inoculated against at baseline. Each measured at follow-up on a 1-7 scale for each of 5 claims, and then summed for a global index (range: 5-35).
Credibility of new claims, exposure #9, follow-up | 2-4 weeks
  Extent to which the claim is credible, extent to which the claim makes you anxious or nervous about the HIV vaccine, likelihood of your sharing the claim, for both HIV vaccine claims specifically inoculated against at baseline. Each measured at follow-up on a 1-7 scale for each of 5 claims, and then summed for a global index (range: 5-35).
Credibility of new claims, exposure #10, follow-up | 2-4 weeks
  Extent to which the claim is credible, extent to which the claim makes you anxious or nervous about the HIV vaccine, likelihood of your sharing the claim, for both HIV vaccine claims specifically inoculated against at baseline. Each measured at follow-up on a 1-7 scale for each of 5 claims, and then summed for a global index (range: 5-35).
Credibility of new claims, exposure #11, follow-up | 2-4 weeks
  Extent to which the claim is credible, extent to which the claim makes you anxious or nervous about the HIV vaccine, likelihood of your sharing the claim, for both HIV vaccine claims specifically inoculated against at baseline. Each measured at follow-up on a 1-7 scale for each of 5 claims, and then summed for a global index (range: 5-35).
Anxiousness o of new claims, exposure #7, follow-up | 2-4 weeks
  Extent to which the claim makes you anxious or nervous about the HIV vaccine for both HIV vaccine claims specifically inoculated against at baseline. Each measured at follow-up on a 1-7 scale for each of 5 claims, and then summed for a global index (range: 5-35).
Anxiousness of new claims, claim #8, follow-up | 2-4 weeks
  Extent to which the claim makes you anxious or nervous about the HIV vaccine for both HIV vaccine claims specifically inoculated against at baseline. Each measured at follow-up on a 1-7 scale for each of 5 claims, and then summed for a global index (range: 5-35).
Anxiousness of new claims, exposure #9, follow-up | 2-4 weeks
  Extent to which the claim makes you anxious or nervous about the HIV vaccine for both HIV vaccine claims specifically inoculated against at baseline. Each measured at follow-up on a 1-7 scale for each of 5 claims, and then summed for a global index (range: 5-35).
Anxiousness of new claims, exposure #10, follow-up | 2-4 weeks
  Extent to which the claim makes you anxious or nervous about the HIV vaccine for both HIV vaccine claims specifically inoculated against at baseline. Each measured at follow-up on a 1-7 scale for each of 5 claims, and then summed for a global index (range: 5-35).
Anxiousness of new claims, exposure #11, follow-up | 2-4 weeks
  Extent to which the claim makes you anxious or nervous about the HIV vaccine for both HIV vaccine claims specifically inoculated against at baseline. Each measured at follow-up on a 1-7 scale for each of 5 claims, and then summed for a global index (range: 5-35).
Shareability of new claims, exposure #7, follow-up | 2-4 weeks
  Likelihood of your sharing the claim, for both HIV vaccine claims specifically inoculated against at baseline. Each measured at follow-up on a 1-7 scale for each of 5 claims, and then summed for a global index (range: 5-35).
Shareability of new claims, exposure #8, follow-up | 2-4 weeks
  Likelihood of your sharing the claim, for both HIV vaccine claims specifically inoculated against at baseline. Each measured at follow-up on a 1-7 scale for each of 5 claims, and then summed for a global index (range: 5-35).
Shareability of new claims, exposure #9, follow-up | 2-4 weeks
  Likelihood of your sharing the claim, for both HIV vaccine claims specifically inoculated against at baseline. Each measured at follow-up on a 1-7 scale for each of 5 claims, and then summed for a global index (range: 5-35).
Shareability of new claims, exposure #10, follow-up | 2-4 weeks
  Likelihood of your sharing the claim, for both HIV vaccine claims specifically inoculated against at baseline. Each measured at follow-up on a 1-7 scale for each of 5 claims, and then summed for a global index (range: 5-35).
Shareability of new claims, exposure #11, follow-up | 2-4 weeks
  Likelihood of your sharing the claim, for both HIV vaccine claims specifically inoculated against at baseline. Each measured at follow-up on a 1-7 scale for each of 5 claims, and then summed for a global index (range: 5-35).

CONTACTS AND LOCATIONS:
Locations (1):
- Health Economics and Epidemiology Research Office, University of the Witwatersrand, Johannesburg, South Africa

IPD SHARING:
Plan to Share IPD: Undecided
The investigators are still determining the data sharing plan and if we will be sharing IPD yet